CLINICAL TRIAL: NCT02617472
Title: Assessment of the Effectiveness of a Pelvic Exercise Device in Strengthening Pelvic Floor Muscles and Treating Urinary Incontinence
Brief Title: Effectiveness of Kegel Exercise Device in Strengthening Pelvic Floor and Treating Urinary Incontinence (UI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lelo Inc. (Industry)
Collaborators: Banner Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT001KSUS
Record Dates: First submitted 2015-10-30; First posted 2015-12-01 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Stress Urinary Incontinence; Sexual Dysfunction
MeSH Terms: conditions — Urinary Incontinence, Stress; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pelvic floor exercise (Experimental): Pelvic floor exerciser, daily use
  Interventions: Device: Pelvic floor exerciser

INTERVENTIONS:
Device: Pelvic floor exerciser — Daily exercise using the study device
  Other Names: KegelSmart pelvic floor trainer

SUMMARY:
This study will assess the effectiveness of a new pelvic floor exercise device in strengthening pelvic floor muscles and treating urinary incontinence among women who are experiencing symptoms of pelvic floor weakness. The study will be conducted over 12 weeks and results will be collected through self-assessment questionnaires and clinical pelvic examination. Effectiveness outcomes will be tracked over the duration of the trial and measured against historical symptoms.

DETAILED DESCRIPTION:
The objective of the study is to test the device with women who are experiencing symptoms of pelvic floor weakness, namely urinary incontinence, vaginal laxity and sexual sensation problems, to assess the changes in pelvic floor muscle strength, before and after the intervention.

The study device is a pelvic floor exercise device that provides biofeedback and exercise guidance.

Women who meet the inclusion criteria will be recruited from the regular patients at the investigation site and given the device to use at home daily for 12 weeks. Subjects will submit information regarding their experience with the device and self-assessed improvements in their symptoms. A pelvic examination will be conducted at the start and conclusion of the study to measure a pelvic floor muscle strength reading.

The research hypothesis is that strength level, subjective assessment of vaginal tightness and sexual sensations will be greater at the end of the study than at the baseline and the mean value of frequency and volume of bladder leaks will be less than at the baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent and HIPAA authorization before any study procedures are conducted;
2. Experience urinary incontinence and/or vaginal laxity and/or decreased sexual sensation for a period of 6 weeks or more.

Exclusion Criteria:

1. Subject has any condition or exhibits behavior that indicates to the Principal Investigator that the Subject is unlikely to be compliant with study procedures and visits
2. Has had prior surgery for incontinence, prolapse or vaginal tightening
3. Has been diagnosed with pelvic organ prolapse more severe than grade 2
4. Suffers from vaginal penetration difficulties
5. Has had more than 3 urinary tract infections in the past 12 months
6. Has any conditions of the bladder that effect continence
7. Suffer from vaginal/vulvar/pelvic pain
8. Is currently taking any medication for incontinence
9. Is pregnant or trying to become pregnant
10. Has given birth less than 6 weeks prior to enrollment
11. Has been diagnosed obese - BMI > 30
12. Is a heavy smoker - > 20 cigarettes per day
13. Has a history of neurological conditions - Parkinson's, multiple sclerosis and other
14. Suffers from chronic constipation

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in pelvic floor strength | 12 weeks
  Pelvic floor strength measured by a clinical perineometer in cm H2O. A baseline measurement of resting and peak muscle contraction values will be recorded at the start before the intervention and after the 12 weeks of treatment.

SECONDARY OUTCOMES:
Frequency of bladder leaks. | 12 weeks
  Reporting of weekly incidence of bladder leaks.
Volume of bladder leaks | 12 weeks
  Reporting of weekly average volume of bladder leaks.A subject assessment with very distinct category gradations.

OTHER OUTCOMES:
Subjective assessment of vaginal tightness | 12 weeks
  Subjective assessment of increased vaginal tone.
Subjective assessment of sexual sensations | 12 weeks
  Subjective assessment based on questions that rate this quality of life parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Wickman, MD, Principal Investigator — FACOG
Locations (1):
- Banner University Medical Center, Phoenix, Arizona, United States